CLINICAL TRIAL: NCT02853448
Title: Evaluation of a Device That Separates Blood Cells From Serum/Plasma for Analysis of Clinical Chemistries
Brief Title: Evaluation of a Device That Separates Blood Cells From Serum/Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H-32418
Record Dates: First submitted 2016-07-27; First posted 2016-08-03 (Estimated); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Plasma Extraction
Keywords: Plasma; Serum; Effective Blood Draws

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Novel Device (Experimental): Every Subject will be assigned to the same arm. This arm calls for blood to be drawn using an original blood drawing apparatus as well as using the novel blood drawing apparatus.
  Interventions: Device: Novel Blood Drawing Apparatus

INTERVENTIONS:
Device: Novel Blood Drawing Apparatus

SUMMARY:
There are many instances where there is no access to a centrifuge (Emergency wards, EMT truck, battle field, etc.) or when a result is needed immediately (myocardial infarction); a new collection tube which could separate serum and plasma from whole blood immediately upon, if not during, collection, would be extremely beneficial. Such a new tube could save time and cost by eliminating centrifugation steps that are currently required to obtain serum and plasma.

DETAILED DESCRIPTION:
A new blood collection tube has recently been developed; the tube separates serum/plasma from the whole blood while the blood flows into the tube. This is accomplished by a filter set inside the tube; the filter set may be impregnated with an anti coagulant agent, such as sodium citrate (blue top) or may be virgin (red top). The serum collection part of the tube is disconnected from the filtering part upon completion of the serum collection, capped with a lid, and forwarded to a bed-side instrument or to a test analysis laboratory. The filter part is discarded in a hazardous waste container. Blood Separation free of red cell damage is achieved by controlling blood flow rate into the device. A 30 second flow intake is typical. The flow rate controller in use in this experiment is an element added in line to the standard blood drawing needle set.

This study is being conducted to compare concentrations of routine clinical chemistries (analytes and electrolytes) measured in serum/plasma obtained from routine standard blood collection tubes to novel blood collection tubes that separate blood cells from whole blood while the blood is being drawn. Routine clinical labs will be performed on the serum and the plasma obtained from the standard and the novel tubes to evaluate the efficacy of the novel tubes to recover cell-free serum for measuring various routine blood analytes as compared to standard tubes.

Procedure Plasma, as well as serum, will be collected and analyzed in the study. While the blood collection procedures for each of these are the same, collection of blood into the standard tube differs from that into the serumSTAT tube; the subsequent post-treatment of the blood/serum/plasma differs from one to the other. The serum will be ready for analysis after completion of the steps. The procedure for how to draw the blood using the new device will be explained and demonstrated to the phlebotomist to ensure (s)he is comfortable using the device.

The following routine clinical chemistry shown in the metabolic panel below shall be measured ;

1. Albumin
2. AlkalinePhosphatase
3. ALT (Alanine Transaminase)
4. AST (Aspartate Transaminase)
5. BUN (Blood Urea Nitrogen)
6. Creatinine
7. Glucose
8. Total Bilirubin
9. Total Protein
10. Calcium
11. Carbon Dioxide
12. Chloride
13. Potassium
14. Sodium
15. Troponin I

Furthermore, the BUN/Creatinine ratio shall also be presented in the data set.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 y/o

Exclusion Criteria:

* NONE

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Number of subjects with similar blood chemistry values for both blood drawing apparatuses | At the time of blood analysis.
  Test analysis will be done between blood chemistry values for both original and novel blood drawing apparatuses. Subject will have blood drawn once, and that blood will be used for a comparative analysis between the two blood drawing apparatuses. Thus, a time frame is N/A in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Holick, MD, PhD, Principal Investigator — Boston University
Locations (1):
- Dr. Solomon Carter Fuller Mental Health Center, 85 E Newton St M-1013, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No